CLINICAL TRIAL: NCT02958319
Title: Clinical Follow-up of Anti-Carbamylated Antibody Status in Rheumatoid Arthritis Patients at 6, 12 and 18 Months
Brief Title: Clinical Follow-up of Anti-Carbamylated Antibody Status in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, David Vega Morales, MD, MsSc, Doctorate, Universidad Autonoma de Nuevo Leon
Other Study IDs: RE16-00001
Record Dates: First submitted 2016-11-02; First posted 2016-11-08 (Estimated); Results first posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: RheumatoId Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Anti P Carb negative RA patients: RA patients negative for antibodies against the carbamylated proteins
- Anti P Carb positive RA patients: RA patients positive for antibodies against the carbamylated proteins

SUMMARY:
Patients with rheumatoid arthritis (RA) with positive antibodies against carbamylated proteins (anti-CarP) have a more severe clinical course. The primary objective of this study in adult subject with RA is as follows: To explore the clinical differences in activity indexes (Disease Activity Score of 28 joints with Erythro Sedimentaion Rate (DAS28-ESR)) at 6, 12 and 18 months of follow up according the anti-CarP antibodies status.

DETAILED DESCRIPTION:
Clinical follow-up of Anti-Carbamylated Antibody Status in Rheumatoid Arthritis patients at 6, 12 and 18 months.

Concept

Patients with rheumatoid arthritis (RA) with positive antibodies against carbamylated proteins (anti-CarP) have a more severe clinical course.

Background

The immune based pathophysiology of RA is one of the most studied. We already know that the citrullinated peptide antigen inducing antibody formation and subsequent anti-cyclic citrullinated peptide (anti-CCP) antibodies. In some patients can explain the clinical manifestations. However it is also apparent that some groups of patients with rheumatoid arthritis who do not have anti-CCP antibodies. It is possible then the presence of a variety of antigens exposed during the disease, and perhaps different clinical presentations associated with each.

The use of anti-CCP antibodies has been included in the classification criteria of RA developed by the American College of Rheumatology (ACR) in 2010 and generated the presence of two sub-groups of patients with RA, the positive and negative for anti-CCP. It is very important to study the presence of anti-CCP antibodies in RA population because it influences the clinical behavior and response to treatment. In very early or undifferentiated arthritis, the presence of anti-CCP antibodies can predict the presence of erosions in the course of the disease. On the other hand, patients with negative anti-CCP antibodies tend to have better responses to treatment with methotrexate.

Initially it was thought that the obvious pathophysiological link between RA and citrullinated peptides leading to formation of antibodies was the apparent cause of the clinical manifestations, but soon it was demonstrated that there were groups of patients with clinical manifestations of RA that did not had anti-CCP antibodies so its genesis was not explained by citrullination. Then it is possible a diversity of antigens exposed during the illness and perhaps different clinical presentations associated with each one or its combinations. So actually, some studies are attempting to show other possible antigens involved in RA and one of them uses homocitrulline as an antigenic basis to RA pathophysiology. The carbamylation or homocitrullination is a posttranslational modification of proteins that occurs when the amino acid lysine reacts with cyanate in a non-enzyme-mediated process generating homocitrulline. Mydel, Bokarewa and cols. demonstrated that immunization of mice with homocitrulline- and citrulline-containing peptides leads to development of erosive arthritis following intra-articular injection of homocitrulline-containing peptides and proposed that homocitrulline induced activation of T cells is a key mechanism in the pathogenesis of autoimmune arthritis as it serves as an initial triggering event for neo-epitope recognition of citrulline containing peptides. Recently It has been shown that rheumatoid arthritis patients has homocitrullinated proteins in his joints which can trigger an inflammatory response with formation of antibodies against homocitrulline.

Shi et al. showed in a study of 571 RA patients and 350 healthy subjects the following statements:

* The anti-carbamylated peptide (Anti-CarP) antibodies are different from Anti-CCP antibodies and they do not cross-react.
* The Anti-CarP antibodies are present in sera of patients with RA.
* Anti-CarP antibodies are found in sera of patients without anti-CCP.
* The Anti-CarP antibodies are associated with increased progression to radiographic damage.

Thus, autoantibodies recognizing anti-CarP are a promising new serological marker for anti CCP antibodies negative RA and are associated with a more severe clinical course.

Hypothesis

Patients with RA with positive antibodies against anti-CarP have a more severe clinical course and elevated cardiovascular risk.

Design

It is a parallel study for clinical follow-up , observational.

Description of Subject Population(s)

* Patients older than 18 years old, both gender, with RA diagnosis according to ACR European Leage Against Rheumatism (EULAR) 2010 classification that accepted and signed informed consent that were seen at the Rheumatology Clinic in Hospital Universitario "Dr. José Eleuterio González", Monterrey, NL. México.
* Exclusion: Chronic kidney disease and pregnant patients Assessment Tools and Procedures
* DAS-28 ESR
* Lipid profile Length of Study in Months
* 18 Primary Endpoints
* Clinical activity measured by DAS28-ESR in patients with RA according to antibodies against anti-CarP status at 6, 12 and 18 months Secondary Endpoints
* Number and accumulative dose of Disease Modifying Anti-Rheumatic Drugs (DMARD) according to antibodies against anti-CarP status at 6, 12 and 18 months
* Cardiovascular risk according to antibodies against anti-CarP status at 6, 12 and 18 months Clinical Information
* Total number of subjects 262
* Number of subjects for each treatment arm 131
* Study Duration Per Patient (in Months) 18

Primary Objective

The primary objective of this study in adult subject with RA is as follows:

1. To explore the clinical differences in activity indexes (DAS28-ESR) at 6, 12 and 18 months of follow up according the anti-CarP antibody status

Study Secondary Objective(s)

One secondary objective is as follows:

* To investigate the remission rate (DAS28-ESR) according the anti-CarP antibody status
* Other secondary objectives are as follows:
* To compare the percentage of subjects with DAS28-ESR Low Disease Activity (LDA) at 6, 12 and 18 months according the anti-CarP antibody status
* To compare the accumulative dose of prednisone between groups according the anti-CarP antibody status
* To compare the number and doses of DMARD´s used to treat RA between groups according the ant CarP antibody status

Study Design

* Prospective, Non-Randomized, Open Label
* Inception Cohort Study

Study Primary Efficacy Endpoints

The primary efficacy endpoitns is as follows:

* The percentage of subjects who meet DAS28-ESR < 2.6 at 6, 12 and 18 months in the Anti CarP positive antibody arm compared Anti CarP negative antibody arm

Study Secondary Efficacy Endpoints

The secondary efficacy endpoints are as follows:

* Percentage of subjects with DAS28-ESR LDA at 6, 12 and 18 months at 6, 12 and 18 months in the Anti CarP positive antibody arm compared Anti CarP negative antibody arm
* Median of the accumulative dose of prednisone at 18 months at 6, 12 and 18 months in the Anti CarP positive antibody arm compared Anti CarP negative antibody arm
* Mean of the number and doses of DMARD´s used to treat RA at enrollment at 6, 12 and 18 months in the Anti CarP positive antibody arm compared Anti CarP negative antibody arm
* Cardiovascular risk according to anti-CarP antibody status

Study Sample Size Calculation

A total of 262 subjects will be followed in this study. According the pilot study it was found a 12 month remission rate in the Anti CarP positive antibody of 33% arm compared Anti CarP negative antibody arm of 50%, with a difference of 17% in remission rate at 12 month follow-up. One hundred and thirty-three patients are needed per group. A 2 group continuity corrected chi square test with a 2-sided significance level (alpha) of 0.05 was used to compare sample size and a 0.2 (beta) to power.

Study Statistical Methods

Descriptive statistic for categorical and numerical variables will be used. Categorical variables will be expressed in frequency and percentage; comparisons will be done by chi square test. Numerical variables, after normality test we will describe them as mean and median with standard deviation (SD) and interquartile range (IQR) as corresponds, respectively.

For the primary end point, chi square test the percentage of DAS28-ESR remission by group will be compared.

For the secondary end points we will compared by t test or Mann Whitnney U the mean o median of the accumulative dose of prednisone and number of DMARD used.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis patients according to ACR EULAR 2010 classification that accepted and signed informed consent

Exclusion Criteria:

* Chronic kidney disease and pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients older than 18 years old, both gender, with RA diagnosis according to ACR EULAR 2010 classification that accepted and signed informed consent that were seen at the Rheumatology Clinic in Hospital Universitario "Dr. José Eleuterio González", Monterrey, NL. México.
  * Exclusion: Chronic kidney disease and pregnant patients
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2016-06; Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Gerardo Garza Leal, PhD, Study Chair — Universidad Autónoma de Nuevo León
Locations (1):
- Servicio de Reumatología, Departamento de Medicina Interna, Facultad de Medicina y Hospital Universitario, Universidad Autonoma de Nuevo León, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
via email request

REFERENCES:
- [Background] Shi J, Knevel R, Suwannalai P, van der Linden MP, Janssen GM, van Veelen PA, Levarht NE, van der Helm-van Mil AH, Cerami A, Huizinga TW, Toes RE, Trouw LA. Autoantibodies recognizing carbamylated proteins are present in sera of patients with rheumatoid arthritis and predict joint damage. Proc Natl Acad Sci U S A. 2011 Oct 18;108(42):17372-7. doi: 10.1073/pnas.1114465108. Epub 2011 Oct 10. PMID 21987802
- [Background] van Venrooij WJ, van Beers JJ, Pruijn GJ. Anti-CCP antibodies: the past, the present and the future. Nat Rev Rheumatol. 2011 Jun 7;7(7):391-8. doi: 10.1038/nrrheum.2011.76. PMID 21647203
- [Background] Turunen S, Koivula MK, Risteli L, Risteli J. Anticitrulline antibodies can be caused by homocitrulline-containing proteins in rabbits. Arthritis Rheum. 2010 Nov;62(11):3345-52. doi: 10.1002/art.27644. PMID 20617522
- [Background] Mydel P, Wang Z, Brisslert M, Hellvard A, Dahlberg LE, Hazen SL, Bokarewa M. Carbamylation-dependent activation of T cells: a novel mechanism in the pathogenesis of autoimmune arthritis. J Immunol. 2010 Jun 15;184(12):6882-90. doi: 10.4049/jimmunol.1000075. Epub 2010 May 19. PMID 20488785
- [Background] Wang Z, Nicholls SJ, Rodriguez ER, Kummu O, Horkko S, Barnard J, Reynolds WF, Topol EJ, DiDonato JA, Hazen SL. Protein carbamylation links inflammation, smoking, uremia and atherogenesis. Nat Med. 2007 Oct;13(10):1176-84. doi: 10.1038/nm1637. Epub 2007 Sep 9. PMID 17828273

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 278 patients were recruited in the study because they fullfilled the four follow-up visits in a retrospective/prospective manner after the informed consent signature and blood sample collection. After antibody analysis, 145 patients were found to be anti-CarP negative and 133 to be anti-CarP positive.
Period: Overall Study
Arm/Group | Anti P Carb Negative RA Patients | Anti P Carb Positive RA Patients
Started | 145 | 133
Completed | 145 | 133
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti P Carb Negative RA Patients | Anti P Carb Positive RA Patients | Total
Number analyzed (Participants) | 145 | 133 | 278
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (11.4) | 55.8 (10.64) | 51.09 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 119 | 254
  Male | 10 | 14 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 145 | 133 | 278
SMOKE [Count of Participants; unit: Participants] | 55 | 59 | 114
DIABETES MELLITUS [Count of Participants; unit: Participants] | 17 | 21 | 38
CARDIOVASCULAR HISTORY [Count of Participants; unit: Participants] | 6 | 3 | 9
HYPERTENSION [Count of Participants; unit: Participants] | 27 | 26 | 53
HYPOTHYROIDSM [Count of Participants; unit: Participants] | 11 | 9 | 20
OSTHEOARTHRITIS [Count of Participants; unit: Participants] | 4 | 4 | 8
FIBROMYALGIA [Count of Participants; unit: Participants] | 3 | 1 | 4
DEPRESSION [Count of Participants; unit: Participants] | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: DAS28-ESR
Description: To explore the clinical differences in activity indexes (DAS28-ESR) at 6, 12 and 18 months of follow-up according the anti-CarP status.
  The DAS28 is a composite score derived from 4 measures, one of them can be the erythrocyte sedimentation rate (ESR). We will be using the DAS28-ESR version. To calculate the DAS28-ESR the rheumatologist or specialist nurse will:- count the number of swollen joints (out of the 28), count the number of tender joints (out of the 28), take blood to measure ESR, ask participants to make a 'global assessment of health' (indicated by marking a 10 cm line between very good and very bad).
  DAS28-ESR is calculated with classic calculators and resulting values are interpreted as follows:
  <2.6: disease remission 2.6 - 3.2: low disease activity 3.2 - 5.1: moderate disease activity >5.1: high disease activity
Time Frame: 6, 12 and 18 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anti P Carb Negative RA Patients | Anti P Carb Positive RA Patients
Number analyzed (Participants) | 145 | 133
units on a scale
  6 MONTHS | 3.75 (1.31) | 3.72 (1.3)
  12 MONTHS | 3.59 (1.46) | 3.69 (1.28)
  18 MONTHS | 3.65 (1.35) | 3.77 (1.32)
Statistical Analysis 1: Comparison: Anti P Carb Negative RA Patients vs Anti P Carb Positive RA Patients; Test type: Superiority; p = 0.82, GENERAL LINEAL MODEL — p < 0.05 was considered statistically significant; GENERAL LINEAL MODEL OF REPEATED MEASURES; Median Difference (Final Values) = 4.1

ADVERSE EVENTS:
Time Frame: 18 MONTHS
Arm/Group | Anti P Carb Negative RA Patients | Anti P Carb Positive RA Patients
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/133
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/133
Other Adverse Events (participants affected / at risk) | 0/145 | 0/133

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT02958319/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT02958319/SAP_001.pdf